CLINICAL TRIAL: NCT03821948
Title: Blood and Stool Sample Collection in Subjects Participating in Colorectal Cancer Screening: Act Bold
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-08
Record Dates: First submitted 2019-01-16; First posted 2019-01-30 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer
Keywords: Blood Draw; Sample Collection; Stool DNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood and stool samples may be used for evaluating performance of biomarkers for feasibility and assay development. Sample may be stored for up to 20 years. These blood and stool samples will be de-identified.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Average CRC Risk Group: Stool sample collection and blood draw in men and women aged 40 and older with average CRC risk undergoing a standard of care colonoscopy procedure
- Increased CRC Risk Group: Stool sample collection and blood draw in men and women aged 40 and older with increased CRC risk undergoing a standard of care colonoscopy procedure

SUMMARY:
The primary objective of this study is to collect de-identified, clinically-characterized stool and whole blood specimens for use in developing and evaluating the performance of new biomarker assays for detection of colorectal cancer (CRC).

DETAILED DESCRIPTION:
Subjects will be men and women, 40 years of age or older who are scheduled for a colonoscopy. Approximately 7,500 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 40 years of age or older.
* Subject is at average or increased risk for development of CRC.
* Subject presents for screening or surveillance colonoscopy.
* Subject has no symptoms that require immediate, or near term, referral for diagnostic or therapeutic colonoscopy.
* Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Any previous cancer diagnosis (with the exceptions of basal cell or squamous cell skin cancers) and/or cancer related treatment (e.g. chemotherapy, immunotherapy, radiation, and/or surgery) within the past 5 years.
* Subject has a diagnosis or personal history of any of the following conditions, including:

  1. Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome).
  2. Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome").
  3. Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis and Familial Hyperplastic Polyposis.
* Subject has a family history of:

  1. Familial adenomatous polyposis (also referred to as "FAP").
  2. Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome").
* Subjects with Cronkhite-Canada Syndrome.
* IV contrast (e.g. CT and MRI) within 1 day [or 24 hours] of blood collection.
* Subject has any condition that in the opinion of the Investigator should preclude participation in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women, 40 years of age or older who are scheduled for a colonoscopy. Approximately 7,500 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5131 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Stool-based biomarkers associated with genetic and epigenetic alterations | Stool sample will be collected prior to initiation of bowel preparation for colonoscopy.
  The outcomes are co-primary. Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in stool from subjects at average risk or increased risk for development of colorectal cancer at the pre-intervention stage.
Blood-based biomarkers associated with genetic and epigenetic alterations. | Point in time blood collection (1 day) at enrollment.
  The outcomes are co-primary. Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood from subjects at average risk or increased risk for development of colorectal cancer at the pre-intervention stage.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - CCT Research/Fiel Family and Sports Medicine, Tempe, Arizona
  - GW Research, Inc, Chula Vista, California
  - Marvel Research, LLC, Huntington Beach, California
  - Desert Medical Group Inc, Palm Springs, California
  - Great Lakes Medical Research, LLC, San Diego, California
  - Connecticut Clinical Research Institute, LLC, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Guardian Angel Research Center, Tampa, Florida
  - DM Clinical Research/Southwest Gastroenterology, Oak Lawn, Illinois
  - Margaret Mary Health, Batesville, Indiana
  - Deaconess Clinic-Mt. Pleasant, Evansville, Indiana
  - Deaconess Clinic-Gateway, Newburgh, Indiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - Capitol Research, Rockville, Maryland
  - Great Lakes Medical Research, LLC, East Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Digestive Disease Care, PC, New Hyde Park, New York
  - Digestive Health Partners, PA, Asheville, North Carolina
  - Charlotte Gastroenterology and Hepatology, LLC, Charlotte, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Great Lakes Medical Research, Beachwood, Ohio
  - Family Practice Center of Wooster, Inc./Clinical Trial Developers, Massillon, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Great Lakes Medical Research, LLC, Westlake, Ohio
  - Comprehensive Internal Medicine, Inc, Wooster, Ohio
  - Great Lakes Medical Research, Erie, Pennsylvania
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Great Lakes Medical Research, LLC, Union City, Tennessee
  - MediSync Clinical Research, Austin, Texas
  - Northside Gastroenterology, Cypress, Texas
  - Vilo Research Group, Inc, Houston, Texas
  - Digestive Health Associates, Houston, Texas
  - DM Clinical Research/PCP For Life, Magnolia, Texas
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Wenatchee Valley Hospital, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures and appendices. The study protocol and informed consent form will also be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will available between 2 and 4 years after publication through the Sponsor.